CLINICAL TRIAL: NCT01268436
Title: Cohort Comparison of Dental Nerve Block With Other Forms of Analgesia in Alleviating the Pain of Toothache
Acronym: Cohort Dental
Status: Completed | Type: Observational
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Wayne Triner, Professor Emergency Medicine, Albany Medical College
Other Study IDs: 2709
Record Dates: First submitted 2010-12-29; First posted 2010-12-30 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2010-12

CONDITIONS: Tooth Pain
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Injectable pain medication: Patients who receive an injectable form of pain medication.
- Oral pain medication: Patients who receive oral pain medication only

SUMMARY:
Toothache is a common source of pain for Emergency Department patients. There are several common ways to control the pain of toothache. But we do not know if any one of them is more effective than another. It is also possible that how we take care of your pain in the Emergency Department will influence the level of pain you experience one or two days from now. This study seeks to answer these questions.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years, pain in any tooth

Exclusion Criteria:

* duration of pain > 96 hours
* oral trauma within 96 hours of presentation
* facial or neck swelling
* pericoronitis
* visual impairment to less than finger counting within three feet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients identified by ED providers as having dental pain will be screened for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2010-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Visual Analog Pain Scale | Before and After treatment of tooth pain
  Is there any change in patient report of pain using the Visual Analog Pain Scale before and after treatment.

SECONDARY OUTCOMES:
Need for additional treatment | while in the Emergency Department
  Does patient require addtional/repeated analgesia or rescue medication?

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center, Albany, New York, United States